CLINICAL TRIAL: NCT02411357
Title: Improving Effective Contraceptive Use Among Opioid-maintained Women: Stage II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Sarah Heil, Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01DA036670 (NIH)
Record Dates: First submitted 2015-04-02; First posted 2015-04-08 (Estimated); Results first posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-01

CONDITIONS: Contraceptive Usage; Opioid Dependence
Keywords: Contraception; Unintended pregnancy; HIV risk; Sexually transmitted infections; Women; Pregnancy; Neonatal health; Drug use; Drug treatment; Opioids
MeSH Terms: conditions — Contraception Behavior; Opioid-Related Disorders; Sexually Transmitted Diseases | interventions — Therapeutics; Fertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment as usual (Active Comparator): The usual care condition will be given general information about contraceptive options and contact information for clinics and providers that provide contraceptive services.
  Interventions: Behavioral: Treatment as usual
- WHO contraception protocol (Experimental): The WHO contraception protocol condition will receive the World Health Organization's contraception protocol and will be invited to attend follow-up visits.
  Interventions: Behavioral: Treatment as usual; Behavioral: WHO contraception protocol
- WHO contraception protocol + incentives (Experimental): The WHO + incentives condition will receive the World Health Organization's contraception protocol and will be invited to attend follow-up visits, but will also receive financial incentives contingent on attending those follow-up visits.
  Interventions: Behavioral: Treatment as usual; Behavioral: WHO contraception protocol; Behavioral: Incentives

INTERVENTIONS:
Behavioral: Treatment as usual — General information about contraceptive options and referral to contraceptive service providers
Behavioral: WHO contraception protocol — World Health Organization's contraception protocol
  Arms: WHO contraception protocol; WHO contraception protocol + incentives
Behavioral: Incentives — Financial incentives contingent on follow-up visit attendance
  Arms: WHO contraception protocol + incentives

SUMMARY:
Nearly 9 of every 10 pregnant opioid-dependent women report that the current pregnancy was unintended and the majority of non-pregnant opioid-maintained women do not use contraception or use less effective methods like condoms. This proposal aims to further test a novel contraceptive management program to increase use of more effective contraceptives among opioid-maintained women at risk of unintended pregnancy.

DETAILED DESCRIPTION:
The rate of unintended pregnancy among opioid-dependent women is extremely high: nearly 9 of every 10 pregnant opioid-dependent women report that the current pregnancy was unintended, a rate 2-3 times that of the general population. Despite these dire statistics, there is a dearth of scientific knowledge about contraceptive use in this population and about how to promote use of more effective contraceptives (e.g., birth control pills, intrauterine devices (IUDs), implants).

The aim of this Stage II Behavioral and Integrative Treatment Development Program application is to further test a novel contraceptive management program to increase use of more effective contraceptives among opioid-maintained (OM) women. OM women at risk for unintended pregnancy (N=195) will be randomly assigned to one of three conditions: (1) usual care, (2) the World Health Organization (WHO) contraception protocol, and (3) the WHO contraception protocol + financial incentives. Participants in the usual care condition will receive a referral to local contraceptive providers. Participants in the WHO alone condition will receive the WHO contraceptive initiation protocol and their choice of prescription contraceptive in consultation with a nurse practitioner. These participants will also subsequently be offered the opportunity to attend 13 follow-up visits where vital signs and a urine pregnancy test will be administered. Side effects of any prescription contraception will also be assessed and participants will have the option to change their prescription contraceptive method at any time. Participants in the WHO + incentives condition will also receive the WHO contraceptive initiation protocol and their choice of prescription contraceptive in consultation with a nurse practitioner. These participants will also subsequently be offered the opportunity to attend 13 follow-up visits where vital signs and a urine pregnancy test will be administered. Side effects of any prescription contraception will be assessed and participants will have the option to change their prescription contraceptive method at any time. Participants in the WHO + incentives condition participants will also earn vouchers exchangeable for goods and services for attending these visits. Contraceptive use by all participants will be evaluated at assessments scheduled 1, 3, 6, and 12 months after trial intake.

ELIGIBILITY:
Inclusion Criteria:

* 18-44 years of age
* pre-menopausal and have no history of tubal ligation or hysterectomy
* have had heterosexual vaginal sex in the past 3 months
* have no plans to become pregnant in the next 6 months
* be medically eligible to use prescription contraceptives
* report no prescription contraceptive use (i.e., no use of pill, patch, ring, implants, or IUDs in the past 7 days or injections in the past 3 months)
* be in opioid maintenance treatment
* at least 8 weeks postpartum
* not be facing imminent incarceration
* have no plans to leave the area in the next 12 months
* be English-speaking

Exclusion Criteria:

* failure to meet the aforementioned inclusion criteria
* refusal to participate

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 138 (Actual)
Dates: Start 2015-05-05 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah H. Heil, Ph.D., Principal Investigator — University of Vermont
Locations (1):
- Vermont Center on Behavior and Health, Burlington, Vermont, United States

REFERENCES:
- [Derived] Heil SH, Melbostad HS, Matusiewicz AK, Rey CN, Badger GJ, Shepard DS, Sigmon SC, MacAfee LK, Higgins ST. Efficacy and Cost-Benefit of Onsite Contraceptive Services With and Without Incentives Among Women With Opioid Use Disorder at High Risk for Unintended Pregnancy: A Randomized Clinical Trial. JAMA Psychiatry. 2021 Oct 1;78(10):1071-1078. doi: 10.1001/jamapsychiatry.2021.1715. PMID 34259798

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: The usual care condition received usual care consisting of a general information brochure about contraceptive methods and contact information for community contraceptive service facilities.
- Contraceptive Services: The contraceptive services condition were offered onsite contraceptive services adapted from the World Health Organization including 6 months of follow-up visits to assess method satisfaction.
- Contraceptive Services + Incentives: The contraceptive services + incentives condition were offered onsite contraceptive services adapted from the World Health Organization including 6 months of follow-up visit to assess method satisfaction plus financial incentives for attending follow-up visits.
Period: Overall Study
Arm/Group | Usual Care | Contraceptive Services | Contraceptive Services + Incentives
Started | 48 | 48 | 42
Completed | 48 | 48 | 42
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Contraceptive Services | Contraceptive Services + Incentives | Total
Number analyzed (Participants) | 48 | 48 | 42 | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.6 (6.0) | 32.0 (5.2) | 31.6 (4.9) | 31.4 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 48 | 42 | 138
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 48 | 48 | 42 | 138
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 1 | 4
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 2 | 1 | 1 | 4
  White | 43 | 45 | 40 | 128
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
One or more unintended pregnancies in lifetime [Count of Participants; unit: Participants] | 41 | 42 | 39 | 122

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Verified Prescription Contraceptive Use at the 6-month Assessment
Time Frame: 6 months after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Contraceptive Services | Contraceptive Services + Incentives
Number analyzed (Participants) | 48 | 48 | 42
Participants | 5 | 14 | 23
Statistical Analysis 1: Comparison: Usual Care vs Contraceptive Services vs Contraceptive Services + Incentives; Test type: Superiority; p < .001, Cochran-Armitage Chi-square trend test

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Usual Care | Contraceptive Services | Contraceptive Services + Incentives
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48 | 0/42
Serious Adverse Events (participants affected / at risk) | 1/48 | 3/48 | 1/42
Other Adverse Events (participants affected / at risk) | 26/48 | 42/48 | 36/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=48) | Contraceptive Services (N=48) | Contraceptive Services + Incentives (N=42)
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Infection secondary to surgical incision (Surgical and medical procedures) | 1 | 0 | 0
Opioid overdose (Psychiatric disorders) | 0 | 1 | 0
Bowel obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Cardiac arrest secondary to probable bupropion overdose (Psychiatric disorders) | 0 | 1 | 0
Hospitalization for depression/suicidality (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=48) | Contraceptive Services (N=48) | Contraceptive Services + Incentives (N=42)
Adverse events not categorized by organ system (General disorders) | 26 (46) | 42 (176) | 36 (230)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/57/NCT02411357/Prot_SAP_000.pdf